CLINICAL TRIAL: NCT01793740
Title: Cognitive Rehabilitation of Children With Sickle Cell Disease: A Pilot Study
Brief Title: Cognitive Rehabilitation in Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00035303
Record Dates: First submitted 2013-02-14; First posted 2013-02-18 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Sickle Cell Disease; Cognitive Impairment
Keywords: sickle cell disease; pediatric; learning disability; cognitive impairment; memory; attention; Children with sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell; Cognitive Dysfunction; Learning Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cogmed (Experimental): These children are enrolled in the Cogmed intervention.
  Interventions: Behavioral: Cogmed
- Waitlist (No Intervention): These children are enrolled in a waitlist condition, after which they will be offered the opportunity to complete the intervention.

INTERVENTIONS:
Behavioral: Cogmed — Computer based program that aims to improve children's memory, attention, and processing speed.
  Other Names: Cogmed computerized cognitive training
  Arms: Cogmed

SUMMARY:
The majority of school-age children with sickle cell disease (SCD) experience neurocognitive deficits, even in the absence of stroke. In particular, deficits in attention and working memory have emerged as two of the most common neurocognitive sequelae of SCD. Thus, the goal of the present proposal is to address feasibility and compliance of a novel computerized cognitive training program, Cogmed. Pilot data will also be collected to establish preliminary efficacy. Twenty-four children meeting initial age and diagnostic criteria will be identified and approached about participation by their attending physician during regularly-scheduled SCD clinic visits. Baseline assessments will include a brief measure of intellectual functioning, a brief cognitive testing battery evaluating processing speed and working memory, in addition to questionnaires regarding behavior and quality of life. Children will then be randomized to the computerized CT program Cogmed (n=12) or a waitlist control (n=12). Participants enrolled in the computerized CT program will be asked to complete 25-sessions of Cogmed over a five to eight week period (3 to 5 sessions per week). Following completion of the program, children and their parents will be asked to return to clinic for a follow-up visit. After a five to eight-week waiting period, children in the waitlist condition will also be asked to return to clinic for a second visit. Following this assessment, participants initially enrolled in the waitlist will be offered an opportunity to participant in the intervention. If interested, they will follow the same intervention protocol described above. These children will return to clinic for a third visit following completion of the intervention. Compliance rate and its confidence interval will be calculated for the overall study population. A t-test for binomial proportion with continuity correction will be used to examine whether the compliance rate is lower than the target. Participants' change in criterion outcomes will be evaluated (i.e., those neurocognitive measures such as attention, executive functioning and working memory, that are most closely related to the trained tasks).

ELIGIBILITY:
Inclusion Criteria:

* 1) Children with a diagnosis of SCD (all genotypes)
* 2) a T-score ≥75th percentile on either the Metacognition or Executive Composite of the BRIEF; and/or
* 3) a standard score ≥1 standard deviation below the mean (<90) on the tasks of executive function or WM from the Cogstate (mean=100; SD=10)

Exclusion Criteria:

* 1) Estimated IQ ≤ 75), or motor, visual, or auditory handicap that prevents computer use;
* 2) a diagnosis of depression or a pervasive developmental disorder (by history);
* 3) clinical stroke (via record medical history); or
* 4) non-English fluency.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2012-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Feasibility | Post-study - Baseline to Post-Intervention, approximately 5 to 8-weeks after baseline assessment
  Feasibility is defined as 75% of subjects completing 80% of the training program.

SECONDARY OUTCOMES:
Efficacy | Baseline to Post-Intervention, approximately 5 to 8-weeks after baseline assessment
  Efficacy will be defined by participant performance on cognitive outcome measures including executive functioning outcomes from the Cogstate.

OTHER OUTCOMES:
Acceptance | After the recruitment period has been completed (approximately 2-years)
  Acceptance is defined by 50% of those approached are able to participate/consent to the study.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie J Bonner, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Child and Family Study Center, Durham, North Carolina, United States